CLINICAL TRIAL: NCT02060773
Title: Effect of EGDT on Hepatic Perfusion in Patients With Septic Shock
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Xiaohua Qiu, physician, Zhongda Hospital
Other Study IDs: zhongdaH
Record Dates: First submitted 2014-02-08; First posted 2014-02-12 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2012-12

CONDITIONS: Septic Shock
Keywords: Septic shock; Early goal directed therapy; Fluid resuscitation; Hepatic perfusion; Indocyanine Green
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To observe the effect of early goal directed therapy (EGDT) on hepatic perfusion in patients with septic shock.

Hypothesis: Hepatic perfusion did not improved after EGDT in patients with septic shock.

DETAILED DESCRIPTION:
Objective To observe the effect of early goal directed therapy (EGDT) on hepatic perfusion in patients with septic shock.

Methods A prospective observational study was carried out. The eligible patients were treated with the standard procedure of EGDT. The hemodynamic data were recorded. Oxygen metabolism and hepatic function were monitored. Indocyanine clearance test was applied to detect the hepatic perfusion. Hemodynamics, hepatic perfusion, oxygen metabolism and hepatic function were compared before treatment, after EGDT and 24 hours after EGDT.

ELIGIBILITY:
Inclusion Criteria:

1. patients with septic shock
2. at least one of the EGDT criteria not achieved
3. informed consent accepted

Exclusion Criteria:

1. ages below 18 or above 90
2. pregnancy
3. the time elapsed over 24 hours after onset of septic shock
4. chronic liver disease
5. terminal stage of disease
6. brain death
7. other types of shock
8. brain injury
9. allergic to iodine or indocyanine

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critical patients with early septic shock admitted to ICU within 24 hours after onset
Sampling Method: Probability Sample
Dates: Start 2012-12; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
ICG-PDR and R15 before treatment, after EGDT and 24 hours after EGDT. | 30 hours

SECONDARY OUTCOMES:
28 days mortality | 28 days
  Follow up to determine the mortality in 28 days after inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Zhongda Hospital of Southeast University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Zhang XW, Xie JF, Liu AR, Huang YZ, Guo FM, Yang CS, Yang Y, Qiu HB. Hepatic Perfusion Alterations in Septic Shock Patients: Impact of Early Goal-directed Therapy. Chin Med J (Engl). 2016 Jul 20;129(14):1666-73. doi: 10.4103/0366-6999.185865. PMID 27411453